CLINICAL TRIAL: NCT02562053
Title: Does Adding Combined Oral Contraceptives to Fluoxetine Improve the Management of Premenstrual Syndrome? A Double Blind Placebo Controlled Study.
Brief Title: Does Adding Oral Contraceptives to Fluoxetine Improve the Management of Premenstrual Syndrome?
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PMS 2
Record Dates: First submitted 2015-09-25; First posted 2015-09-29 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Premenstrual Syndrome
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Fluoxetine; Contraceptives, Oral, Combined

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fluoxetine (Active Comparator): Women will receive daily oral fluoxetine 20 mg in addition to an oral placebo similar to COC daily for 21 days starting from the 3rd day of menstruation.
  Interventions: Drug: Fluoxetine; Drug: Placebo 1
- Combined oral contraceptives and fluoxetine (Active Comparator): Women will receive COC containing drospirenone (drospirenone 3mg+Ethinylestradiol 0.03mg; Yasmin® Schering AG, Egypt) daily for 21 days starting from the 3rd day of menstruation in addition to oral fluoxetine 20 mg daily.
  Interventions: Drug: Fluoxetine; Drug: Combined oral contraceptives
- Placebo (Placebo Comparator): Women will receive oral placebo similar to COC daily for 21 days starting from the 3rd day of menstruation in addition to a daily oral placebo similar in size, color and structure to fluoxetine
  Interventions: Drug: Placebo 1; Drug: Placebo 2

INTERVENTIONS:
Drug: Fluoxetine — Women will receive oral fluoxetine 20 mg daily.
  Arms: Combined oral contraceptives and fluoxetine; Fluoxetine
Drug: Combined oral contraceptives — women will receive COC containing drospirenone (drospirenone 3mg+Ethinylestradiol 0.03mg; Yasmin® Schering AG, Egypt) daily for 21 days starting from the 3rd day of menstruation
  Arms: Combined oral contraceptives and fluoxetine
Drug: Placebo 1 — Women will receive oral placebo similar to COC daily for 21 days starting from the 3rd day of menstruation
  Arms: Fluoxetine; Placebo
Drug: Placebo 2 — Women will receive a daily oral placebo similar to fluoxetine
  Arms: Placebo

SUMMARY:
Three hundred women with severe premenstrual syndrome will be divided into 3 groups using computer generated random numbers. Group 1 will receiveCombined oral contraceptives (COC) containing drospirenone (drospirenone 3mg+Ethinylestradiol 0.03mg) daily for 21 days starting from the 3rd day of menstruation in addition to oral fluoxetine 20 mg daily. Group 2 will receive fluoxetine 20 mg daily in addition to an oral placebo similar to COC daily for 21 days starting from the 3rd day of menstruation.Group 3 will receive oral placebo similar to COC daily for 21 days starting from the 3rd day of menstruation in addition to a daily oral placebo similar in size, color and structure to fluoxetine.

DETAILED DESCRIPTION:
Premenstrual syndrome (PMS) manifests with distressing physical, behavioral and psychological symptoms, in the absence of organic or underlying psychiatric disease, which regularly recur during luteal phase of each menstrual cycle and disappear or significantly improve by the end of menstruation. Approximately 85-90 % of women may experience premenstrual emotional and physical changes in their reproductive age and the prevalence of severe PMS ranges from 3% to 8%.

The etiology of PMS is unknown but cyclical ovarian activity and the effect of estradiol and progesterone on serotonin and gamma-amino butyric acid are key factors. Absence of PMS before puberty, in pregnancy and after the menopause supports a role of cyclical ovarian activity in PMS etiology. PMS symptoms include psychological symptoms like mood swings, irritability, depression and feeling out of control; physical symptoms like breast tenderness, bloating and headaches; and behavioral symptoms like reduced visuospatial and cognitive ability. To diagnose PMS, symptoms should be recorded prospectively over two cycles using a symptom diary. Several symptom diaries exist but the Daily Record of Severity of Problems (DRSP) is reliable, simple for patients and recommended by the Royal College of Obstetricians and Gynecologists.

Life style modifications like stress reduction, exercise, and low carbohydrate diet have been suggested for management of PMS but have not been thoroughly investigated. Pharmacological treatments of PMS include COC, serotonin reuptake inhibitors gonadotrophin-releasing hormone agonists, anxiolytics, and diuretics. Various other treatments have also been recommended including acupuncture, dietary supplements, and bright light therapy, PMS treatment should be based on individual symptoms, concomitant medical history and the need of contraception.

The objective of the study is to investigate the role of the combined use of fluoxetine and COC versus fluoxetine in the treatment of PMS.

Three hundred women with severe premenstrual syndrome will be divided into 3 groups using computer generated random numbers. Group 1 will receive COC containing drospirenone (drospirenone 3mg+Ethinylestradiol 0.03mg) daily for 21 days starting from the 3rd day of menstruation in addition to oral fluoxetine 20 mg daily. Group 2 will receive fluoxetine 20 mg daily in addition to an oral placebo similar to COC daily for 21 days starting from the 3rd day of menstruation.Group 3 will receive oral placebo similar to COC daily for 21 days starting from the 3rd day of menstruation in addition to a daily oral placebo similar in size, color and structure to fluoxetine.

To diagnose PMS women will be asked to document their symptoms daily for 2 months using the daily record of severity of problems (DRSP). DRSP is a questionnaire comprised of 25 physical and emotional symptoms including impairment of physical and social activities, women will be asked to give a score of 1 to 6 for each symptom 1 = not at all, 2 = minimal, 3 = mild, 4 = moderate, 5 = severe, 6 = extreme. The investigators will add the symptoms scores of the first day of menses and PMS will be excluded if the score is< 50. If the total score is greater than 50, the investigators will recorded two cycles of symptoms. If more than three items have an average score of more than 3 (mild) during the luteal phase, the investigators will add the scores of five-day intervals during the luteal and follicular phases. PMS will be diagnosed when the luteal phase score is 30 percent greater than the follicular phase score in the 2 months. All women will have a psychiatric review and women with underlying psychiatric disease will be excluded. Women who are unable to interact socially or professionally because of the symptoms will be considered to have severe PMS. All married women will be advised to use barrier contraceptives.

All women will be asked to take the medications for 6 months and record their symptoms using the DRSP. Women with suboptimal social or professional interaction will be considered having moderate PMS. Women with no interference with the social or professional activity will be considered as having mild PMS. Women with day 1 DRSP score <50 and women with average luteal phase scores <30% more than the average proliferative scores will not be considered having PMS.

ELIGIBILITY:
Inclusion Criteria:

* Severe PMS
* Regular periods

Exclusion Criteria:

* Underlying psychiatric disease.
* Body mass index > 35.
* Women on combined oral contraceptives.
* History of deep venous thrombosis, known liver, kidney or heart disease.
* Allergy to COC or fluoxetine

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Improved PMS | Monthly for 6 months.
  Women will be asked to document their symptoms daily using DRSP. Cured PMS will be diagnosed if day 1 DRSP score is< 50 or if the luteal phase score is not at least 30 percent greater than the follicular phase score.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - BeniSuef University hospitals, BeniSuef
  - Cairo University Hospitals, Cairo

REFERENCES:
- [Background] Marjoribanks J, Brown J, O'Brien PM, Wyatt K. Selective serotonin reuptake inhibitors for premenstrual syndrome. Cochrane Database Syst Rev. 2013 Jun 7;2013(6):CD001396. doi: 10.1002/14651858.CD001396.pub3. PMID 23744611
- [Background] Yonkers KA. Management strategies for PMS/PMDD. J Fam Pract. 2004 Sep;Suppl:S15-20. No abstract available. PMID 15508358
- [Background] Steiner M, Brown E, Trzepacz P, Dillon J, Berger C, Carter D, Reid R, Stewart D. Fluoxetine improves functional work capacity in women with premenstrual dysphoric disorder. Arch Womens Ment Health. 2003 Feb;6(1):71-7. doi: 10.1007/s00737-002-0162-2. PMID 12715267
- [Background] Lopez LM, Kaptein AA, Helmerhorst FM. Oral contraceptives containing drospirenone for premenstrual syndrome. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD006586. doi: 10.1002/14651858.CD006586.pub4. PMID 22336820